CLINICAL TRIAL: NCT04091958
Title: Reconstruction of Partial Mastectomy Defects With Myo-glandular Local Flap: Pilot Study.
Brief Title: Reconstruction of Partial Mastectomy Defects With Pectoralis Myo-glandular Local Flap.
Status: Unknown | Phase: Phase 1 | Type: Interventional
Last Known Status: Recruiting
Sponsor: Mansoura University (Other)
Responsible Party: Principal Investigator, Osama Hussein, Professor of Surgery, Mansoura University
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: R/19.08.578
Record Dates: First submitted 2019-09-13; First posted 2019-09-17 (Actual); Last update posted 2020-11-19 (Actual); Status verified 2020-11

CONDITIONS: Breast Cancer
Keywords: Breast conserving surgery; Pectoralis major muscle
MeSH Terms: conditions — Breast Neoplasms

STUDY DESIGN:
Intervention Model Description: This is a cohort study.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Post-tumourectomy reconstruction with myo-glandular flap. (Experimental): Standard tumourectomy followed by reconstruction with myo-glandular flap.
  Interventions: Procedure: Pectoralis myo-glandular flap reconstruction.

INTERVENTIONS:
Procedure: Pectoralis myo-glandular flap reconstruction. — Tumorectomy with surgical margin will be evaluated with frozen-section examination. Reconstruction starts with mobilization of skin flaps. The sternal head of the pectoralis major muscle will be disconnected from its insertion at the humerus. The muscle fibers will be mobilized off the chest wall. The pectoralis major receives dual blood supply. The pectoral branches of the thoraco-acromial artery enter the superior part of the muscle and the perforator branches of the internal mammary artery enter the medial part of the muscle. According to the location of the defect in the breast, the muscle will be mobilized based on one vascular pedicle. The muscle flap may consist of all or some segmental fibres of the sternal head of the pectoralis major muscle. In all cases, the muscle flap connection to the overlying breast parenchyma is kept intact and the clavicular head of the pectoralis major muscle is undisturbed. Closure of the cavity in layers over suction drain will follow.

SUMMARY:
Increasing number of breast cancer patients are being treated with conservative surgery; without the need for mastectomy. The cosmetic sequel of breast conservative surgery can be unsatisfactory to the patient and may necessitate secondary surgery. The present study aims at improving the cosmetic outcome of breast conservative surgery. The defect remaining in the breast tissue after excision of the tumour will be filled with the underlying pectoralis major muscle. This pilot study will test the safety and efficacy of using the pectoralis major muscle for reconstructing a partial mastectomy defect. fifteen patients with early breast cancer scheduled for breast conservation will be recruited to this study.

DETAILED DESCRIPTION:
Breast conservative surgery is the standard of care for early breast cancer patients. Large multi-center randomized trials have shown breast conservative surgery to be non-inferior to total mastectomy . Oncoplastic breast surgery consists of adequate tumorectomy followed by aesthetic repair of the partial mastectomy defect to achieve satisfactory cosmetic outcome. Oncoplastic surgery is recommended for all breast conservative operations. Level-I oncoplastic surgery is used to repair minor loss of breast volume. In this level, reconstruction is limited to mobilization and redistribution of the breast parenchyma to fill the tumorectomy defect. Larger volume loss requires complex procedures with significant morbidity and is called level-II oncoplasty. In level-II procedures, extra-mammary tissue is mobilized to fill the breast defect (volume replacement). Alternatively, bilateral reduction mammoplasty procedure (volume displacement) is used to reconfigure the breast, obliterate the tumorectomy defect and correct associated breast hypertrophy or ptosis. With either strategy, volume replacement and volume displacement require extensive skin incisions and tissue mobilization. Thus, level-II oncoplasty achieve maximum aesthetic outcome on the expense of major surgical trauma and significant probability of operative morbidity. Recent years have witnessed renewed interest in de-escalating oncoplastic surgical strategies. Level-I oncoplastic operations have been used more frequently to fulfil the cosmetic needs of the majority of breast conservative operations. Moreover, the patient acceptability of the complex level-II oncoplastic procedures is not universal. With the exception of level-II oncoplastic procedures, breast cancer surgery is a well-tolerated intervention that can be offered in a fast-track or day-case basis with economic, psychological and social advantages.

In view of the above-mentioned considerations, The investigators and others have worked to expand the role of level-I oncoplastic surgery. Several innovative techniques have been recommended to allow repair of wider post-tumorectomy defects with simple mobilization of breast parenchymal flaps.

The pectoralis major muscle flap is the classic workhorse of reconstructive surgery of the head and neck. The muscle has been extensively used as a pedicled or free flap to achieve reconstruction of major post-ablative tissue defects. In aesthetic breast surgery, pectoralis major muscle has been used as a sling to correct breast ptosis.

The investigators hypothesized that mobilization of glandular tissue based on underlying pectoralis major fibres will allow repair of larger defects using an "extended level-I oncoplasty". Pectoralis major is known to have reliable segmental blood supply that allows muscle-sparing flap construction with minimal or no functional deficit.

The aim of this work is to evaluate the operative and aesthetic outcome of extended-level-I oncoplastic reconstruction with pectoralis myo-parenchymal flaps.

This is a pilot study that is equivalent to a phase I trial i.e. a safety study. The primary goal is to identify unforeseen surgical, oncologic or cosmetic drawbacks for the technique. This study will also evaluate the efficacy of the technique for providing satisfactory cosmetic outcome.

ELIGIBILITY:
Inclusion Criteria:

1. Patients with early breast cancer or phylloides tumor.
2. Eligible for breast conservative surgery.
3. Expected post-lumpectomy volume loss of 20-40% of breast volume.
4. Tumor location in upper quadrants.
5. Informed consent.

Exclusion Criteria:

1. Patient refusal.
2. Contraindication of breast conservative therapy:

   1. Pregnancy.
   2. Diffuse microcalcifications.
   3. Patient choice for mastectomy.
   4. Collagen / vascular disease.
   5. Multicentric tumor.
3. Psychological co-morbidity.

Min Age: 18 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 15 (Estimated)
Dates: Start 2019-08-24 (Actual); Primary Completion 2021-01-30 (Estimated); Study Completion 2022-02-28 (Estimated)

PRIMARY OUTCOMES:
The rate of major complications | Six weeks after surgery.
  The rate of major complications related to surgery that necessitate further intervention.
The score of early cosmetic outcome | Six weeks after surgery.
  This is a categorical variable. The cosmetic score is reported according to the Harris method. In this method the overall cosmetic result is ranked as one of four scores. The maximum score is "Excellent" where the treated breast is identical to the other breast. Slight difference is scored as "Good". Marked difference without distortion is scored as " Fair". The least score is " Poor" where there is breast distortion.

SECONDARY OUTCOMES:
The score of late cosmetic outcome | 12 Months after surgery.
  This is a categorical variable. The cosmetic score is reported according to the Harris method. In this method the overall cosmetic result is ranked as one of four scores. The maximum score is "Excellent" where the treated breast is identical to the other breast. Slight difference is scored as "Good". Marked difference without distortion is scored as " Fair". The least score is " Poor" where there is breast distortion.

OTHER OUTCOMES:
The percentage of adequate resection | Two weeks after surgery.
  This variable is dichotomous. Histopathological examination of the paraffin blocks of the resected tumour specimen will be used to describe the resection safety margin. The safety margin will be scored as either adequate or inadequate. Adequate safety margin indicates no tumor on inked surface of the resected specimen. Inadequate safety margin indicates presence of tumour on inked surface of the resected specimen.

CONTACTS AND LOCATIONS:
Overall Officials: Osama Hussein, MD,PhD.FEBS, Principal Investigator — Mansoura University
Locations (1):
- Mansoura University Oncology Center, Al Mansurah, DK, Egypt

IPD SHARING:
Plan to Share IPD: Undecided

REFERENCES:
- [Background] Harris JR, Levene MB, Svensson G, Hellman S. Analysis of cosmetic results following primary radiation therapy for stages I and II carcinoma of the breast. Int J Radiat Oncol Biol Phys. 1979 Feb;5(2):257-61. doi: 10.1016/0360-3016(79)90729-6. No abstract available. PMID 110740
- [Background] Tobin GR. Pectoralis major segmental anatomy and segmentally split pectoralis major flaps. Plast Reconstr Surg. 1985 Jun;75(6):814-24. doi: 10.1097/00006534-198506000-00009. PMID 4001201
- [Background] Fisher B, Anderson S, Bryant J, Margolese RG, Deutsch M, Fisher ER, Jeong JH, Wolmark N. Twenty-year follow-up of a randomized trial comparing total mastectomy, lumpectomy, and lumpectomy plus irradiation for the treatment of invasive breast cancer. N Engl J Med. 2002 Oct 17;347(16):1233-41. doi: 10.1056/NEJMoa022152. PMID 12393820